CLINICAL TRIAL: NCT04268706
Title: A Phase 2 Multi-Center Study Evaluating the Safety and Efficacy of CD30-Directed Genetically Modified Autologous T Cells (CD30.CAR-T) in Adult and Pediatric Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Phase 2 Study Evaluating Autologous CD30.CAR-T Cells in Patients With Relapsed/Refractory Hodgkin Lymphoma (CHARIOT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tessa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESSCAR001
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin Lymphoma, Adult; Hodgkin Disease Recurrent; Hodgkin Disease Refractory; Hodgkin Disease, Pediatric
Keywords: r/r Hodgkin Lymphoma, CD30, adult, pediatrics
MeSH Terms: conditions — Hodgkin Disease | interventions — fludarabine; fludarabine phosphate; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD30 positive r/r classical Hodgkin Lymphoma (Experimental): Patients with relapsed or refractory classical Hodgkin Lymphoma who have failed 3 prior lines of treatment, which may include a prior autologous and/or allogeneic stem cell transplant.
  Patients will be treated with autologous CD30.CAR-T cells.
  Interventions: Drug: CD30.CAR-T; Drug: Fludarabine; Drug: Bendamustine

INTERVENTIONS:
Drug: CD30.CAR-T — Autologous CD30.CAR-T cells infused on Day 0 after the completion of lymphodepleting chemotherapy.
Drug: Fludarabine — Lymphodepletion chemotherapy (30 mg/m2/day) for 3 consecutive days
  Other Names: Fludara
Drug: Bendamustine — Lymphodepletion chemotherapy (70 mg/m2/day) for 3 consecutive days
  Other Names: Bendeka

SUMMARY:
This is a two-part, Phase 2, multicenter, open-label, single arm study to evaluate the safety and efficacy of autologous CD30.CAR-T in adult and pediatric subjects with relapsed or refractory CD30+ classical Hodgkin Lymphoma.

DETAILED DESCRIPTION:
The Pilot part of the study will evaluate the safety, tolerability, and preliminary antitumor efficacy of CD30.CAR-T. The Pivotal part of the study will evaluate antitumor efficacy and further evaluate safety and tolerability. All study eligibility requirements, assessments, procedures, and follow-up are the same for patients in both Pilot and Pivotal parts of the study.

Subjects who meet eligibility criteria will have their blood drawn by leukapheresis for manufacture the CD30.CAR-T cells. Subjects are allowed bridging chemotherapy, as per Investigator choice, while waiting for production of CD30.CAR-T. Lymphodepletion (LD) with fludarabine and bendamustine will be administered for 3 consecutive days starting on Day -5 to Day -3, prior to CD30.CAR-T infusion, which will be administered on Day 0 as a single IV infusion. Depending on disease status, eligible subjects may receive up to a total of two CD30.CAR-T infusions at the same dose, each with preceding LD chemotherapy.

Subjects will be closely monitored for safety and efficacy throughout the Treatment Period until the end of study (EOS) visit at Month 24. Subjects will be followed for survival, withdrawal of consent or study closure, whichever occurs first. Health Related Quality of Life assessments will also be collected throughout the study. After the EOS visit, subjects will enter the long-term follow-up phase (LTFU) which will include survival follow-up, additional safety, efficacy and biomarker assessments, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is determined prior to blood collection . Patients must satisfy the following criteria to be enrolled in the study:

1. Signed Informed Consent Form
2. Male or female patients who are 12 - 75 years of age
3. Histologically confirmed classical Hodgkin Lymphoma
4. Relapsed or refractory cHL that has failed at least 3 prior lines of therapy, including:

   * chemotherapy
   * BV and/or
   * PD-1 inhibitor Patients may have previously received an autologous and/or allogeneic stem cell transplant
5. CD30-positive tumor
6. At least 1 measurable lesion according to The Lugano Classification
7. Laboratory parameters: Hematological, renal and hepatic functions, and coagulation parameters

   * Hgb ≥ 8.0 g/dL
   * Total bilirubin ≤ 1.5 × ULN
   * AST and ALT ≤ 5 × the ULN
   * CrCl > 45 mL/min
   * ANC >1,000/µL
   * Platelets >75,000/µL
   * PT or INR ≤ 1.5 × ULN; PTT or aPTT ≤ 1.5 × ULN
8. ECOG PS of 0 to 1 or equivalent [either Karnofsky PS (for patients ≥ 16 year of age) or Lansky PS (for patients < 16 years of age)]
9. Anticipated life expectancy > 12 weeks

Exclusion Criteria:

1. Evidence of lymphomatous involvement of central nervous system (CNS)
2. Presence of clinically relevant or active seizure disorder, stroke, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement
3. Active uncontrolled bleeding or a known bleeding diathesis
4. Inadequate pulmonary function defined as pulse oximetry < 90% on room air
5. ECHO or MUGA with LVEF < 45%
6. On-going treatment with immunosuppressive drugs or chronic systemic corticosteroids
7. Having received:

   * Anti-CD30 antibody-based therapy within 4 weeks prior to CD30.CAR-T infusion
   * Prior investigational CD30.CAR-T
   * CD30 bispecific agent within 8 weeks prior to CD30.CAR-T infusion
   * Autologous HSCT within 90 days or allogeneic HSCT within 180 days prior to CD30.CAR-T infusion
8. Currently receiving any investigational agents within 4 weeks prior to study enrollment; or received any tumor vaccines within 6 weeks prior to CD30.CAR-T infusion
9. Active acute or chronic graft versus host disease (GVHD) requiring immune suppression regardless of grade
10. Evidence of human immunodeficiency virus (HIV) infection
11. Seropositive for and with evidence of active viral infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
12. Unresolved > Grade 1 non-hematologic toxicity associated with any prior treatments
13. History of hypersensitivity reactions to murine protein-containing products or other product excipients
14. Symptomatic cardiovascular disease: Class III or IV according to the New York Heart Association (NYHA) Functional Classification
15. Active second malignancy or history of another malignancy within the last 3 years
16. Women who are pregnant or intending to become pregnant; women who are breastfeeding; persons with procreative potential not using and not willing to use 2 highly effective methods of contraception
17. Any other serious, life-threatening, or unstable preexisting medical conditions

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2037-03 (Estimated)

PRIMARY OUTCOMES:
Pilot: Safety of autologous CD30.CAR-T | Minimum 24 months post-CD30.CAR-T infusion
  Adverse events
Pivotal: Anti-tumor effect of autologous CD30.CAR-T using objective response rate (ORR) as assessed by an Independent Radiology Review Committee (IRRC) per the Revised Criteria for Response Assessment: The Lugano Classification (Cheson, 2014) | As early as 6 weeks after CD30.CAR-T treatment
  ORR

SECONDARY OUTCOMES:
Pilot: Antitumor efficacy of autologous CD30.CAR-T using objective response rate (ORR) as assessed by an Independent Radiology Review Committee (IRRC) per the Revised Criteria for Response Assessment: The Lugano Classification (Cheson et al., 2014) | As early as 6 weeks after CD30.CAR-T treatment
  ORR
Pilot: Duration of Response | Minimum 24 months post-CD30.CAR-T infusion
  DOR
Pilot: Progression Free Survival | Minimum 24 months post-CD30.CAR-T infusion
  PFS
Pilot: Overall Survival | Minimum 24 months post-CD30.CAR-T infusion
  OS
Pilot: Health Related quality of life (HRQoL) questionnaire | Minimum 24 months post-CD30.CAR-T infusion
  QoL
Pivotal: Number of patients with adverse events as a measure of safety and tolerability of CD30.CART cells | As early as 6 weeks after CD30.CAR-T treatment
  Adverse events
Pivotal: Objective response rate (ORR as assessed by IRRC) per the Revised Criteria for Response Assessment: The Lugano Classification (Cheson, 2014) | Minimum 24 months post-CD30.CAR-T infusion
  ORR
Pivotal: Progression Free Survival (PFS) | Minimum 24 months post-CD30.CAR-T infusion
  PFS
Pivotal: Duration of Response (DOR) | Minimum 24 months post-CD30.CAR-T infusion
  DOR
Pivotal: Overall Survival | Minimum 24 months post-CD30.CAR-T infusion
  OS
Pivotal: Health Related quality of life (HRQoL) questionnaire | Minimum 24 months post-CD30.CAR-T infusion
  HRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No